CLINICAL TRIAL: NCT04749004
Title: Healthy.Tyrol - A Randomized-Controlled Lifestyle Intervention to Increase Physical Activity Levels in Adolescents
Brief Title: A Randomized-Controlled Lifestyle Intervention to Increase Physical Activity Levels in Adolescents
Acronym: healthy tyrol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VASCage GmbH (Other)
Collaborators: Management Center Innsbruck (Unknown); Medical University Innsbruck (Other); Tirol Kiniken GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: healthy.tyrol
Record Dates: First submitted 2020-09-23; First posted 2021-02-10 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Life Style, Healthy; Life Style
Keywords: Lifestyle Intervention; Adolescents; Health Behavior; Financial Incentives; Commitment Contract; Nudges; Cardiovascular Risk Reduction; Primoridal Prevention; Physical Activity
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Tracking of steps by means of a fitness tracker
  For the economic experiments on time and risk preferences monetary rewards are used with the amount depending on the decisions of the participants.
  Participants collect points for transmitting informations about the amount of steps taken on the basis of which they get a small reward (e.g., a skiing ticket)
  Setting-up of a commitment contract on the individual's goal of monthly steps taken
  Provision of financial incentives upon achievement of one's goal of steps taken
  Provision of nudges (reminders)
  Interventions: Behavioral: Promotion of physical activity
- Control Group (No Intervention): Tracking of steps by means of a fitness tracker
  For the economic experiments on time and risk preferences monetary rewards are used with the amount depending on the decisions of the participants.
  Participants collect points for transmitting informations about the amount of steps taken on the basis of which they get a small reward (e.g., a skiing ticket)
  To keep incentives constant the control group will also receive the flat payment of €10 to disentangle the effects between the contract and financial incentives.

INTERVENTIONS:
Behavioral: Promotion of physical activity — Provision of motivational stimuli (commitment contracts, nudges, financial incentives) to increase amount of steps taken
  Arms: Intervention Group

SUMMARY:
Students at the age of 14-16 years will be randomized to one intervention arm or one control arm in a 1:1 ratio. Participants of both groups receive a fitness tracker to count the amount of their steps taken. The participants of the intervention arm will commit themselves to a personal goal of steps taken by means of a commitment contract. Achievement of the goal will be rewarded with financial incentives to fulfill the requirements of proper reward medium, according to the Induced Value Theory (Smith, 1976).

The duration of the intervention will be 1 year; incentives are provided for 6 months, the remaining 6 months are the follow-up period.

The hypothesis is that intensified motivational strategies like the provision of commitment contracts and nudges are effective in increasing the number of steps taken per month compared to a control group.

DETAILED DESCRIPTION:
Adolescents age 14 to 16 years visiting schools throughout Tyrol, Austria will be randomized to one intervention arm or a control arm on a class-wise level in a 1:1 ratio. Participants will be invited by the Department of Education in Tyrol and schools will be contacted directly. At the baseline examination cardiovascular risk profiles (including laboratory analysis; anthropometry; a standardized medical interview; and blood pressure, bioelectrical impedance and pulse-wave velocity measurements) are determined and results are communicated in an individual discussion of results.

Afterwards, participants of both groups receive a fitness tracker to count the amount of their steps taken. The participants of the intervention arm will commit themselves to a personal goal of steps taken by means of a commitment contract. Achievement of the goal will be rewarded with financial incentives to fulfill the requirements of proper reward medium, according to the Induced Value Theory (Smith, 1976) and nudges (reminders) will be provided to increase motivation.

The duration of the intervention will be 1 year; incentives are provided for 6 months, the remaining 6 months are the follow-up period. After 1 year a follow-up examination will be conducted. Economic experiments on time and risk preferences are furthermore carried out at baseline.

The hypothesis is that intensified motivational strategies like the provision of commitment contracts and nudges are effective in increasing the number of steps taken per month compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 - 16 years at baseline
* Signed informed consent of subjects and legal guardian

Exclusion Criteria:

* Persons, who are suspended upon a court order or upon other legal processes or are accommodated according to the Hospitalization Act, or for whom a custodian is appointed (or appointment is initiated).
* Persons with impaired power of judgment
* Persons who are currently engaged in military or community service

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 373 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Difference in average number of steps taken per day | month 1 versus months 2-7
  Baseline (observation period = first month) versus intervention period (months 2-7)

SECONDARY OUTCOMES:
Difference in average number of steps taken per day | month 1 versus month 8 to follow-up examination
  Baseline (observation period = first month) versus post-intervention period (month 8 - follow-up examination)
Achievement of pre-defined goal of steps (specified as percentage change compared to baseline; 0-50% increase) | month 1 versus months 2-7
  percentage of participants in the intervention group achieving their predefined goal (using explanatory variables such as demographic variables, time and risk preferences etc.
Difference in number of ideal cardiovascular health metrics in the ideal range as defined by the American Heart Association | 15 months
  Between and within group differences
Difference in average minutes of moderate to vigorous physical activity per day | 15 months
  Between and within group differences
Difference in systolic and diastolic blood pressure | 15 months
  Between and within group differences
Difference in body composition as measured by bioeletrical impedance | 15 months
  Between and within group differences
Magnitude of commitment (specified as as percentage increase of steps taken by steps of 10 percentage points ranging from 0% - 50%) | 15 months
  Between group differences
Difference in visceral abdominal fat-tissue thickness as measured by ultrasonography | 15 months
  Between and within group differences
Difference in liver fat and fibrosis as measured by FibroScan | 15 months
  Between and within group differences Liver fat content is assessed by means of the Controlled-Attenuation Parameter [dB/m] and fibrosis by means of transient elastography [kPa].
Predictors of progression of Intima-Media Thickness [µm] | 15 months
  Intima-media thickness is assessed by means of ultrasonography, predictors to be examined include: Blood pressure, lipid parameters, age, sex, liver fat and fibrosis, body composition/BMI, smoking, fasting glucose and CRP.
Predictors of progression of pulse-wave velocity [m/s] | 15 months
  pulse-wave velocity is measured using the Vicorder, an oscillometric pulse-wave velocity measurement device, predictors to be examined include: Blood pressure, lipid parameters, age, sex, liver fat and fibrosis, body composition/BMI, smoking, fasting glucose and CRP.

OTHER OUTCOMES:
The role of time and risk preferences on long-term habit formation (of physical activity in amount of steps taken). | 15 months
  Time and risk preferences are assessed by means of economic experiments specific for each preference, steps taken are assessed by means of a fitness tracker/step counter.
The role of time and risk preferences on the change of the amount of steps taken per day every month during the motivation period and afterwards in comparison to the baseline value at month 1 | 15 months
  Time and risk preferences are assessed by means of economic experiments specific for each preference, steps taken are assessed by means of a fitness tracker/step counter.
The impact of physical activity on primary headache disorders. | 15 months
  Physical acitivity is assessed by means of a fitness tracker (with step counting function) and by structured physician-guided interviews. Primary headache disorders are assessed in structured physician-guided interviews and classified according to the ICHD-3. Parameters include frequency, intensity, duration, headache characteristics and concomitant symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knoflach, MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No